CLINICAL TRIAL: NCT04132804
Title: Pilot Study Investigating the Effect of Tai Chi as Treatment for IBS-C
Brief Title: Effect of Tai Chi as Treatment for IBS-C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Kyle Staller, MD, MPH, Assistant Professor in Medicine, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019P000361
Record Dates: First submitted 2019-08-21; First posted 2019-10-21 (Actual); Results first posted 2021-10-29 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Irritable Bowel Syndrome With Constipation
MeSH Terms: interventions — Tai Ji

STUDY DESIGN:
Intervention Model Description: This is a single-center pilot study. All patients enrolled in the study will participate in the Tai Chi treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tai Chi Treatment (Experimental): All patients in the trial will receive 1-hour Tai Chi lessons once per week for a total of 8 weeks.
  Interventions: Behavioral: Tai Chi

INTERVENTIONS:
Behavioral: Tai Chi — Tai Chi Chuan (taijiquan) or Tai Chi is a mind-body practice borne of Chinese philosophy and martial arts which has been practiced for centuries to promote deep relaxation, strengthened health, and to prevent injuries and illness.

SUMMARY:
The purpose of the study is to evaluate the efficacy of Tai Chi practice in reducing symptoms of Irritable Bowel Syndrome with Constipation (IBS-C).

DETAILED DESCRIPTION:
This is a single-center pilot study investigating the efficacy of Tai Chi practice in reducing symptoms of IBS. The investigators hope that subjects practicing Tai Chi will have reduced symptoms of IBS-C as measured through overall global symptom relief as well as the IBS-SSS, IBS-QOL, VSI, HADS, Visual Analogue Pain Scale, and changes in bloating, abdominal pain, abdominal distention, and constipation severity. The study will also use daily entries made through the GeoPain app to record trends in pain intensity.

ELIGIBILITY:
Inclusion

1. Age 18 - 70 years
2. BMI ≤ 35
3. Rome IV criteria for IBS-C
4. Continued IBS-C throughout run-in period
5. Compliant with reporting during run-in
6. Ability to follow verbal and written instructions
7. Ability to record daily patient reported outcomes via RedCap survey
8. Ability to use the GeoPain app on a smart phone
9. Ability to use Zoom as a platform for conducting study visits virtually
10. Ability to respond to 80% of the daily diaries
11. Ability to attend at least 7 out of 8 Tai Chi classes
12. Informed consent form signed by the subjects

Exclusion

1. Unwilling to abstain from participation in Tai Chi (other than that provided for the study) or other mind-body practices (i.e. yoga that is new to regimen) until completion of the study
2. Non-English speaking
3. Participation in any other clinical trial with active intervention within the last 30 days
4. Non-compliance with reporting during run-in period
5. Inability to stand without assistance for 20 minutes
6. Patients reporting any usage of a prohibited medication during the run-in period
7. History of regular opiate or narcotic pain-reliever use
8. Current use of prescribed or illicit opioids
9. Change in current medication regimen related to GI motility, laxatives, or antidepressants
10. Abdominal pain severity of 4 on a 0-4 visual analogue scale, where 4 is the worst possible pain, during pre-screen or run-in
11. Severe osteoarthritis
12. Severe rheumatoid arthritis
13. Severe constipation defined as <1 bowel movement per week without use of laxatives
14. History of GI lumen surgery (including gastric bypass) at any time or other GI or abdominal operations within 60 days prior to entry into the study
15. History of small bowel resection (except if related to appendectomy)
16. Subjects anticipating surgical intervention during the study
17. Angina, coronary bypass, or myocardial infarction within 6 months prior to Screening Visit
18. Crohn's disease or ulcerative colitis
19. History of intestinal stricture (e.g., Crohn's disease)
20. BMI >35
21. Pregnancy (or positive urine pregnancy test(s) in females of childbearing potential)
22. Known history of diabetes (type 1 or 2)
23. History of gastroparesis
24. History of abdominal radiation treatment
25. History of pancreatitis
26. History of malabsorption or celiac disease
27. History of intestinal obstruction or subjects at high risk of intestinal obstruction including suspected small bowel adhesions
28. History of human immunodeficiency virus
29. History of cancer within the past 5 years (except adequately-treated localized basal cell skin cancer or in situ uterine cervical cancer)
30. Neurological disorders, metabolic disorders, or other significant disease that would impair their ability to participate in the study
31. Any other clinically significant disease interfering with the assessments according to the Investigator (e.g., disease requiring corrective treatment, potentially leading to study discontinuation)
32. Any relevant biochemical abnormality interfering with the assessments according to the Investigator
33. Inability to attend at least 7 out of the 8 Tai Chi classes
34. Inability to respond to 80% of the daily diaries

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2022-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Staller, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tai Chi Treatment
Started | 31
Completed | 20
Not Completed | 11

BASELINE CHARACTERISTICS:
Arm/Group | Tai Chi Treatment
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (15.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 3
  Black or African American | 1
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 31
Body Mass Index, kg/m^2 [Mean (Standard Deviation); unit: kg/m^2] | 23.4 (4.6)
Waist circumference, cm [Mean (Standard Deviation); unit: cm] | 85.4 (10.9)
IBS Symptom Severity Score [Mean (Standard Deviation); unit: score on a scale] | 232.8 (110.3)
Hospital Anxiety and Depression Score [Mean (Standard Deviation); unit: score on a scale] | 15.1 (6.1)
IBS Quality of Life Score [Mean (Standard Deviation); unit: score on a scale] | 91.0 (31.5)
Visceral Sensitivity Index Score [Mean (Standard Deviation); unit: score on a scale] | 48.4 (17.8)
Visual Analogue Abdominal Pain Scale Score [Mean (Standard Deviation); unit: score on a scale] | 1.8 (0.8)
Bowel movement frequency [Mean (Standard Deviation); unit: movements per day] | 1.4 (1.1)
Constipation severity [Mean (Standard Deviation); unit: score on a scale] | 3.4 (2.6)
Abdominal discomfort severity [Mean (Standard Deviation); unit: score on a scale] | 4.3 (2.3)
Bloating severity [Mean (Standard Deviation); unit: score on a scale] | 5.0 (2.3)
Global Assessment of Relief [Mean (Standard Deviation); unit: score on a scale] | 3.4 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: IBS Symptom Severity Score at 12 Weeks
Description: Questionnaire involves yes/no questions, entering numbers, rating scales from 0 to 100, and marking locations of pain. No subscales. Total score is derived by multiplying the number of days of pain (0 to 10) by 10 and summing it with the value from each of 4 scales (0 to 100). Higher total score represents greater symptom severity (min score= 0, max score= 500).
Time Frame: At final study visit, 12 weeks.
Population: Patients who completed the study in its entirety.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tai Chi Treatment
Number analyzed (Participants) | 20
score on a scale | 184.7 (99.2)

2. Secondary Outcome: Likelihood of Continuing Treatment
Description: A 5-point scale indicating likelihood of continuing Tai Chi as a treatment where 1 represents least likelihood and 5 represents greatest likelihood.
Time Frame: Recorded at final study visit (following 8 weeks of treatment)
Population: Patients who completed the study in its entirety.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tai Chi Treatment
Number analyzed (Participants) | 20
score on a scale | 4.2 (1.1)

3. Secondary Outcome: Treatment Satisfaction
Description: A 5-point scale indicating satisfaction with Tai Chi treatment where 1 represents the least satisfaction and 5 represents the most satisfaction
Time Frame: Recorded at final study visit (following 8 weeks of treatment)
Population: Patients who completed the study in its entirety.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tai Chi Treatment
Number analyzed (Participants) | 20
score on a scale | 4 (0.9)

4. Secondary Outcome: IBS Quality of Life (IBS-QOL) at 12 Weeks
Description: Questionnaire about the quality of life of those with IBS. All questions rated from 1 to 5. Higher ratings represent worse quality of life. Subscales exist for dysphoria, interference with activity, body image, health worry, food avoidance, social reaction, sexual, and relationship. Subscales are summed for the total composite score. Primary interest in this study will be the total composite score. Higher total composite score represents greater symptom severity (min score= 34, max score= 170).
Time Frame: At final study visit, 12 weeks
Population: Patients who completed the study in its entirety.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tai Chi Treatment
Number analyzed (Participants) | 20
score on a scale | 79.8 (33.5)

5. Secondary Outcome: Daily Bowel Movement Frequency at 12 Weeks
Description: Number of complete spontaneous bowel movements (csbm) per week. Bowel movements reported daily. Reported outcome is mean number of bowel movements reported at the final study visit.
Time Frame: At final study visit, 12 weeks.
Population: Patients who completed the study in its entirety.
Measure: Mean (Standard Deviation); unit: movements per day
Arm/Group | Tai Chi Treatment
Number analyzed (Participants) | 20
movements per day | 1.4 (0.8)

6. Secondary Outcome: Bloating Scale Score at 12 Weeks
Description: A 10-point scale indicating bloating severity where 0 represents the least severity and 10 represents the most severity.
Time Frame: At final study visit, 12 weeks
Population: Patients who completed the study in its entirety.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tai Chi Treatment
Number analyzed (Participants) | 20
score on a scale | 4.1 (2.9)

7. Secondary Outcome: Abdominal Discomfort Scale Score at 12 Weeks
Description: A 10-point scale indicating abdominal discomfort severity where 0 represents the least severity and 10 represents the most severity.
Time Frame: At final study visit, 12 weeks.
Population: Patients who completed the study in its entirety.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tai Chi Treatment
Number analyzed (Participants) | 20
score on a scale | 3.3 (2.7)

8. Secondary Outcome: Constipation Severity Scale Score at 12 Weeks
Description: A 10-point scale indicating constipation severity where 0 represents the least severity and 10 represents the most severity.
Time Frame: At final study visit, 12 weeks.
Population: Patients who completed the study in its entirety.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tai Chi Treatment
Number analyzed (Participants) | 20
score on a scale | 3.4 (3.1)

9. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS) Score at 12 Weeks
Description: Questionnaire about depression and anxiety severity. All questions rated from 0 to 3. Higher ratings represent greater severity. Subscales exist for depression and anxiety. Subscales are summed for the total composite score. Higher scores represents greater severity (min score= 0, max score= 21 for both subscales; min score= 0, max score= 42 for total score).
Time Frame: At final study visit, 12 weeks.
Population: Patients who completed the study in its entirety.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tai Chi Treatment
Number analyzed (Participants) | 20
score on a scale | 13.3 (8.0)

10. Secondary Outcome: Visceral Sensitivity Index (VSI) Score at 12 Weeks
Description: Questionnaire about visceral sensitivity severity. All questions rated from 1 to 6. Higher ratings represent greater severity. No subscales. Scores for questions are summed for a total score. Higher total score represents greater symptom severity (min score= 15, max score= 90).
Time Frame: At final study visit, 12 weeks
Population: Patients who completed the study in its entirety.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tai Chi Treatment
Number analyzed (Participants) | 20
score on a scale | 53.6 (19.4)

11. Secondary Outcome: Stool Microbiome
Description: Difference in microbiome (presence, absence, abundance, diversity) before treatment (baseline) versus after treatment.
  Pan-microbial (bacterial, archaeal, viral, and eukaryotic) taxonomic profiles will be determined using MetaPhlAn2 which identifies taxa to the strain level and quantifies their relative abundances. Functional genomic profiles, detailed species-specific reconstruction of microbial metabolic pathways, their complement of gene orthologs, taxonomic distributions, and abundances will be generated with HUMAnN2, providing taxon-specific profiles of gene families and pathways to survey microbial community metabolic potential in each metagenome.
  Intestinal contents appear different from person to person in terms of microbial presence therefore we do not have a specific list of microbes that will be assessed.
  Microbe diversity will be measured in relative abundance. Data have not yet been reported as funding has not been acquired for this level of analysis at this time.
Time Frame: Change from baseline to final visit. Through study completion, up to 18 weeks
Reporting Status: Not Posted, anticipated posting 2022-12

12. Secondary Outcome: Global Assessment of Relief at 12 Weeks
Description: A 7-point scale indicating overall IBS symptom relief where 1 represents completely relieved and 7 represents completely worse.
Time Frame: At final study visit, 12 weeks
Population: Patients who completed the study in its entirety.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tai Chi Treatment
Number analyzed (Participants) | 20
score on a scale | 3.4 (0.9)

ADVERSE EVENTS:
Time Frame: The time over which each participant was assessed was 14 weeks. This time frame includes 2 weeks of run-in screening, 8 weeks of Tai Chi treatment, and 4 weeks of follow-up.
Arm/Group | Tai Chi Treatment
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 1/31
Other Adverse Events (participants affected / at risk) | 0/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tai Chi Treatment (N=31)
Serious (Gastrointestinal disorders) | 1 (1) — Emergency Room visit as recommended by provider for evaluation of SBO due to no BM in 8 days, and subsequent discharge same day. Subject ceased participation in the study during the 2 week run-in period. SAE occurred prior to intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-22): https://cdn.clinicaltrials.gov/large-docs/04/NCT04132804/Prot_SAP_000.pdf